CLINICAL TRIAL: NCT01873105
Title: The CARS Study: Communicating About Readiness (for Discharge)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Froedtert Hospital (Other)
Responsible Party: Principal Investigator, Marianne Weiss, Associate Professor, Marquette University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PRO00019092
Record Dates: First submitted 2013-04-26; First posted 2013-06-07 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Hospital Discharge Communication Processes

STUDY DESIGN:
Intervention Model Description: Before/after implementation of a health team communication intervention. 2 samples.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health team educational intervention (Experimental): Agency for Healthcare Research and Quality (AHRQ) TeamSTEPPS approach will be used to redesign health team communication processes regarding preparation for discharge. This redesign will be followed by education for all health team members.
  Interventions: Other: Health Team Educational Intervention
- Control pre-intervention (No Intervention): Usual care control before implementation of the health team communication intervention

INTERVENTIONS:
Other: Health Team Educational Intervention — AHRQ TeamStepps processes will be used to redesign health team discharge communication processes and an educational intervention for health care team members
  Arms: Health team educational intervention

SUMMARY:
The purpose of this study is to improve the experience of discharge of adult medical surgical patients through improved discharge preparation communication between patients and care team members, with subsequent improvement in the post-discharge experience. Obtaining multiple perspectives on discharge readiness creates the opportunity for patient and care team to partner in identifying deficiencies in discharge readiness that warrant anticipatory, compensatory, or corrective interventions prior to discharge, with the goal of averting post-discharge problems and utilization. The results will also inform development and translation of tools for assessment of discharge readiness to clinical care environments.

DETAILED DESCRIPTION:
Specific Aims are to:

1. Describe patterns of communication about discharge and collaboration among members of the health care team
2. Conduct psychometric testing of 3 forms of the Readiness for Hospital Discharge Scale (RHDS - MD, RN, Patient)
3. Describe relationships between care team communication, patient perceptions of quality of discharge preparation and perceived readiness for discharge, care team (RN and MD) assessments of discharge readiness, and post-discharge outcome ( post-discharge coping difficulty, Emergency Department (ED) use, and 30 day readmission.
4. Determine the impact of an intervention with the inpatient care team to improve discharge preparation communication.

H1: Patient perceptions of discharge readiness, post-discharge coping difficulty, ED use and readmission will improve following a care team educational intervention about discharge preparation, compared to pre-intervention baseline measures.

H2: Care team members will report improved frequency and amount of discharge preparation communication following a care team educational intervention about discharge preparation, compared to pre-intervention baseline measures.

H3: RN-MD collaboration will increase following a care team educational intervention about discharge preparation, compared to pre-intervention baseline measures

ELIGIBILITY:
Inclusion Criteria:

* inpatient care team members from 2 nursing units of an academic medical center: Attending physician, resident, medical students, mid-level providers, staff RNs, and case managers/discharge coordinators
* adult medical-surgical patients admitted the 2 nursing units who are at least 18 years of age, speak English, and discharged directly home

Exclusion Criteria:

* patient discharged home with hospice care
* patients not discharged directly home
* decisionally incapacitated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Readmission | 30 days post discharge
  Readmission within the 30 days after hospital discharge
Emergency Department visits | 30 days post discharge
  ED visits within the 30 days after hospital discharge

SECONDARY OUTCOMES:
Post-discharge Coping Difficulty Scale | 14 to 21 days post-hospitalization
  Coping difficulty after hospital discharge measured using the Post-Discharge Coping Difficulty Scale is collected via telephone followup between 14 and 21 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Weiss, DNSc RN, Principal Investigator — Marquette Unoversity; Kristi Opper, MS RN, Principal Investigator — Froedtert Hospital
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States